CLINICAL TRIAL: NCT04654286
Title: Clinical Outcomes of Human Amniotic Membrane and Allogeneic Mesenchymal Stem Cells Composite Augmentation for Nerve Transfer Procedure in Brachial Plexus Injury Patients
Brief Title: Human Amniotic Membrane and Mesenchymal Stem Cells Composite
Acronym: BPI+MSC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Soetomo General Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 647 / Panke.KKE/ XI / 2016
Record Dates: First submitted 2020-11-18; First posted 2020-12-04 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-11

CONDITIONS: Brachial Plexus Neuropathies
Keywords: Brachial Plexus Injury; Amniotic Membrane; Mesenchymal Stem Cells; Nerve Transfer
MeSH Terms: conditions — Brachial Plexus Neuropathies | interventions — Nerve Transfer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Nerve transfer procedure) (Active Comparator): Patient will receive nerve transfer procedure without augmentation
  Interventions: Procedure: Nerve transfer procedure
- Experimental group (Nerve transfer with HAM-AdMSC composite wrapping) (Experimental): Following nerve transfer procedure, the end-to-end anastomosis will be wrapped with HAM-AdMSC composite as augmentation
  Interventions: Procedure: Nerve transfer with HAM-AdMSC composite wrapping

INTERVENTIONS:
Procedure: Nerve transfer procedure — 1. Identification of potential donor nerves: phrenic nerve, accessory nerve, intercostal nerve, motor branch nerve innervating long head of triceps muscle, motor branch of ulnar nerve innervating flexor carpi ulnaris (FCU) muscle, and motor branch of median nerve innervating flexor carpi radialis (FCR) muscle.
  2. Donor nerve is checked for its viability with an electric stimulator during surgery
  3. Viable donor nerve is dissected, transferred to the recipient area, and sutured with end-to-end anastomosis.
  Arms: Control group (Nerve transfer procedure)
Procedure: Nerve transfer with HAM-AdMSC composite wrapping — When the nerve transfer procedure is finished, the end-to-end anastomosis is wrapped by a composite consisted of human amniotic membrane and allogeneic adipose-derived mesenchymal stem cells (HAM-AdMSC)
  Arms: Experimental group (Nerve transfer with HAM-AdMSC composite wrapping)

SUMMARY:
The purpose of this clinical trial is to investigate the utility of composite wrapping comprising human amniotic membrane and allogeneic adipose-derived mesenchymal stem cells (HAM-AdMSC) for augmentation of nerve transfer procedure in upper TBPI patients

DETAILED DESCRIPTION:
Nerve transfer procedure is recognized as the current gold standard for treating traumatic brachial plexus injury (TBPI). However, despite the current major progress in diagnosis and microsurgical repair, the prognosis in TBPI remains unfavorable due to limited donor nerve and compromised regenerative capability of the nervous system arising from prolonged denervation. Therefore, there is a major need to devise new treatment strategies; and one possible approach is to develop cellular therapies to bioengineer new nerve tissue and/or modulate the endogenous regenerative mechanisms within the injured nerve.

Our previous studies have shown that the peripheral nerve tissue engineering approach using human amniotic membrane seeded with allogeneic adipose-derived MSCs to augment axonal regeneration in nerve transfer of TBPI patient revealed promising functional recovery of the shoulder range of motion (ROM). The investigators plan a non-randomized clinical trial in a single center to investigate the use of a hybrid (composite) between human amniotic membrane (HAM) and allogeneic adipose-derived mesenchymal stem cells (AdMSC) as wrapping in the nerve transfer procedure of upper TBPI patients, with a focus on the augmentation of axonal regeneration

ELIGIBILITY:
Inclusion Criteria:

* Suffering from upper BPI (C5-C6 and/or C5-C7) for a duration of fewer than 12 months
* Have no systemic disease (Diabetes Mellitus, Lupus erythematosus, rheumatoid arthritis)
* Without prior medicamentous treatment history such as corticosteroids
* Agree to contribute in the study

Exclusion Criteria:

* Complete BPI (C5-Th1), lower BPI (C8-Th1)
* Traumatic BPI associated with delayed/non-union fracture of the upper extremity affected side.
* Polytrauma conditions which are not fully recovered

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-11-17 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Active range of motion (AROM) pre-surgery | Pre-surgery
  Shoulder: flexion, extension, abduction, adduction, external rotation, internal rotation. Elbow: flexion and extension. Forearm: pronation and supination. The tests are performed by two blinded assessor, and expressed in degrees.
Active range of motion (AROM) at 12 months follow-up | 12 months
  Shoulder: flexion, extension, abduction, adduction, external rotation, internal rotation. Elbow: flexion and extension. Forearm: pronation and supination. The tests are performed by two blinded assessor, and expressed in degrees.
Functional motor power outcome pre-surgery | Pre-surgery
  Measured by Medical Research Council (MRC) scale. The MRC scale consists of 6 values of motor power evaluation, ranging from 0 to 5 (0=No contraction, 1=Flicker or trace contraction, 2=Active movement but eliminated with gravity, 3=Active movement against gravity, 4=Active movement against gravity and resistance, 5=Normal power). The tests are performed by two blinded assessor. A higher score indicates better functional motor power outcome.
Functional motor power outcome at 12 months follow-up | 12 months
  Measured by Medical Research Council (MRC) scale. The MRC scale consists of 6 values of motor power evaluation, ranging from 0 to 5 (0=No contraction, 1=Flicker or trace contraction, 2=Active movement but eliminated with gravity, 3=Active movement against gravity, 4=Active movement against gravity and resistance, 5=Normal power). The tests are performed by two blinded assessor. A higher score indicates better functional motor power outcome.

SECONDARY OUTCOMES:
Initial elbow flexion MRC grade 1 (in months) | throughout the study duration (12 months), recorded as the first time reported by the patients
  Measurement of the length of time (in months) for the patients to show initial contraction (achieve MRC grade 1) of elbow flexion. Previous study by Estrella (2011) showed that the average time for brachial plexus injury patients to achieve an elbow flexion grade M3 after nerve transfer procedure was 7.6 months (range, 5-12 months). As the elbow flexion is the most important movement to restore in treating BPI, the investigators aim to compare the length of time (in months) for the patients to achieve initial contraction (MRC grade 1). The sooner the patients achieve initial elbow flexion MRC grade 1, the better the outcome is.
Initial elbow flexion MRC grade 3 (in months) | throughout the study duration (12 months), recorded as the first time reported by the patients
  Measurement of the length of time (in months) for the patients to achieve MRC grade 3 (active movement against gravity) of elbow flexion. Previous study by Estrella (2011) showed that the average time for brachial plexus injury patients to achieve an elbow flexion grade M3 after nerve transfer procedure was 7.6 months (range, 5-12 months). As the elbow flexion is the most important movement to restore in treating BPI, the investigators aim to compare the length of time (in months) for the patients to achieve MRC grade 3. The sooner the patients achieve initial elbow flexion MRC grade 3, the better the outcome is.
Pain outcome pre-surgery | Pre-surgery
  Measured by visual analogue scales (VAS). Patients are asked to described their level of pain from the scale 0 to 10 (0 indicating no pain, 1-3 indicating mild pain, 4-6 indicating moderate pain, 7-9 indicating severe pain, and 10 indicating worst, unbearable pain). The lower scores mean a better pain outcome.
Pain outcome at 12 months follow-up | 12 months
  Measured by visual analogue scales (VAS). Patients are asked to described their level of pain from the scale 0 to 10 (0 indicating no pain, 1-3 indicating mild pain, 4-6 indicating moderate pain, 7-9 indicating severe pain, and 10 indicating the worst, unbearable pain). The lower scores mean a better pain outcome.
Disabilities of the Arm, Shoulder, and Hand (DASH) score pre-surgery | pre-surgery
  DASH score is a self-assessment of symptoms and function of the entire upper extremity comprising 30 items. Each item consists of five levels of answers (1=no difficulty/symptoms, 2=mild difficulty/symptoms, 3=moderate difficulty/symptoms, 4=severe difficulty/symptoms, and 5=extreme difficulty (unable to do)/symptoms). The scores are then used to calculate a scale score ranging from 0 (no disability) to 100 (most severe disability). Greater DASH scores reflect greater disability (worse outcome).
Disabilities of the Arm, Shoulder, and Hand (DASH) score at 12 months follow-up | 12 months
  DASH score is a self-assessment of symptoms and function of the entire upper extremity comprising 30 items. Each item consists of five levels of answers (1=no difficulty/symptoms, 2=mild difficulty/symptoms, 3=moderate difficulty/symptoms, 4=severe difficulty/symptoms, and 5=extreme difficulty (unable to do)/symptoms). The scores are then used to calculate a scale score ranging from 0 (no disability) to 100 (most severe disability). Greater DASH scores reflect greater disability (worse outcome).
Short Form-36 (SF-36) score pre-surgery | pre-surgery
  A generic, multipurpose, short-form health survey comparing the relative burden of diseases consisting of 36 questions which cover eight domains of health namely physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. Each domain is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. A higher score indicating a more favourable health state/quality of life (better outcome).
Short Form-36 (SF-36) score at 12 months follow-up | 12 months
  A generic, multipurpose, short-form health survey comparing the relative burden of diseases consisting of 36 questions which cover eight domains of health namely physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. Each domain is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. A higher score indicating a more favourable health state/quality of life (better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Heri Suroto, MD,PhD, Principal Investigator — Dr. Soetomo General Academic Hospital/ Universitas Airlangga
Locations (1):
- Cell and Tissue Bank - Regenerative Medicine, Dr. Soetomo General Academic Hospital/ Faculty of Medicine Universitas Airlangga, Surabaya, East Java, Indonesia